CLINICAL TRIAL: NCT06384053
Title: Skin Cancer and Hyperthermia and Radiotherapy - SAHARA a Two-arm, Open-label, Randomized Controlled Phase II Trial
Brief Title: Skin Cancer and Hyperthermia and Radiotherapy
Acronym: SAHARA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Winterthur KSW (Other)
Collaborators: Luzerner Kantonsspital (Other); Lindenhofgruppe AG (Industry); Kantonsspital Aarau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHARA Trial
Record Dates: First submitted 2024-04-15; First posted 2024-04-25 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-01

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma Skin; Non-melanoma Skin Cancer
Keywords: BCC; SCC skin; w-IRA hyperthermia; radiotherapy for non-melanoma skin cancer; non-melanoma Skin cancer; w-IRA combined with RT; hyperthermia
MeSH Terms: conditions — Carcinoma, Basal Cell; Hyperthermia | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperthermia -Experimental Group A (Experimental): The study arm in which hyperthermia and radiotherapy are administered. The RT Dose: 6 fractions of 5 Gy each, delivered twice per week and with a minimum interval of 48 hours, preferably 72 hours, between each fraction over three weeks.
  Interventions: Combination Product: Water-filtered infrared-A-hyperthermia (wIRA) hyperthermia combined; Radiation: Radiotherapy (RT)
- Radiotherapy - Control Group (Active Comparator): The study arm in which only radiotherapy is administered. RT Dose: 12 fractions of 4 Gy each, delivered 3 times per week, with sessions scheduled every other day (exceptions can be made in weeks with holidays) over four weeks.
  Interventions: Radiation: Radiotherapy (RT)

INTERVENTIONS:
Combination Product: Water-filtered infrared-A-hyperthermia (wIRA) hyperthermia combined — The wIRA device applies hyperthermia by heating the treatment area (with maximum surface temperature set to 43° C), aiming to make cancer cells more sensitive to radiation therapy for non-melanoma skin cancer combined with radiotherapy.
  Arms: Hyperthermia -Experimental Group A
Radiation: Radiotherapy (RT) — Radiotherapy is applied.

SUMMARY:
The SAHARA trial assesses wether combining ultrahypofractionated accelerated radiotherapy (RT) with hyperthermia is as effective as standard hypofractionated high-dose radiation in treating non-melanoma skin cancer (NMSC).

DETAILED DESCRIPTION:
The SAHARA Trial is investigating if adding hyperthermia to radiotherapy (RT) can enhance treatment outcomes by making cancer cells more sensitive to radiation, thus requiring lower doses and potentially reducing side effects. The trial compares high-dose RT alone with de-escalated RT plus hyperthermia. The aim is to demonstrate that the combination is non-inferior to standard RT in treating non-melanoma skin cancer (NMSC). The trial is designed for elderly people of 65 years or older.

ELIGIBILITY:
Inclusion Criteria:

* Personally signed and dated written informed consent
* Histologically confirmed invasive non-melanoma skin cancer (NMSC), including basal cell carcinoma (BCC) and squamous cell carcinoma (SCC) of any differentiation
* ≥ T2 (TNM Classification 8th Edition)
* Tumor thickness up to 2cm (Maximum Depth invasion and/or exophytic growth, measured on pathology report or imaging)
* Local recurrence allowed, if primary treatment longer ago than 6 months (after primary treatment other than radiotherapy (RT))
* Age ≥ 65 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2, with a life expectancy of more than 6 months
* Presentation at the Swiss Hyperthermia Network (SHN) tumor conference mandatory

Exclusion Criteria:

* Other histology than BCC or SCC
* T1 tumor and/or N+ (according to TNM classification 8th edition)
* Tumors after resection (R1 or R2 as well as adjuvant indication)
* Tumor invasion into critical areas
* Several lesions exceeding the capacity of one treatment/radiation field (multiple lesions within one treatment field are acceptable)
* Previous (one month) or concurrent Chemo- or Immunotherapy
* Patients with connective tissue disorders (e.g. Sclerodermia, Lupus erythematodes)
* Lesions inside or in proximity (within 3cm) previously irradiated area
* Medical immunosuppression
* wIRA-specific exclusion criteria

  * Tattoos in irradiated area
  * Increased photosensitivity (either due to simultaneous treatment with photosensitivity-enhancing medications or conditions such as porphyria)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Local control | Within two years post-treatment initiation.
  The primary outcome is local control, defined as the absence of of recurrence or need for subsequent intervention.

SECONDARY OUTCOMES:
Analysis | Immediately (within 24 hours post-treatment), at six weeks post-treatment and at three months post-treatment.
  Radiation is applied assessed immediately post-treatment, at six weeks, and three months post-treatment using Common Terminology Criteria for Adverse events (CTCAE 5.0).
Late toxicities | at 6months, one year and two years post-treatment
  Monitoring late toxicities, specifically noted at six months, one year, and two years after completion of treatment using Common Terminology Criteria for Adverse events (CTCAE 5.0).
Quality of life assessment | at three months, 6months, one year and two years post-treatment
  Evaluations are carried out at time of inclusion, immediately post-treatment, at three months, 6months, one year and two years post-treatment utilizing the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire for Elderly (QLQ-ELD14) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Arnold, Dr.med.univ.(A), Principal Investigator — Luzerner Kantonsspital; Maximilian Sturz, Dr.med., Principal Investigator — Luzerner Kantonsspital
Locations (4):
- Switzerland (4):
  - Kantonsspital Aarau, Aarau, Canton of Aargau
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - Lindenhofgruppe, Bern
  - Luzerner Kantonsspital, Lucerne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arnold W, Sturz M, Batifi N, Vaupel P, Notter M, Mueller-Hubenthal B, Puric E, Brodmann S, Zwahlen D. Skin cancer and hyperthermia and radiotherapy - SAHARA: study protocol for a multicenter, two-arm, open-label, randomized controlled phase II non-inferiority trial. Trials. 2025 Dec 22;26(1):574. doi: 10.1186/s13063-025-09274-y. PMID 41430304